CLINICAL TRIAL: NCT05379023
Title: Integrating Home-Based Video Teleneuropsychology Into Clinical Practice: Typical Versus Atypical Alzheimer's Disease
Brief Title: VIdeo Telehealth in ALzheimer's: NeuroPsychology (VITAL-NP)
Acronym: VITAL-NP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: 21-5037; R21AG072153 (NIH)
Record Dates: First submitted 2022-05-02; First posted 2022-05-18 (Actual); Results first posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Suspected Typical Alzheimer's Disease (AD); Suspected Atypical Alzheimer's Disease (AD)

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Face-to-face evaluation (FF), TeleNP evaluation (Other): In-Person (standard of care) Modality completed first, Telehealth Modality completed second
  Interventions: Behavioral: Face-to-face evaluation (FF); Behavioral: TeleNP evaluation
- TeleNP evaluation, Face-to-face evaluation (FF) (Other): Telehealth Modality completed first, In-Person (standard of care) Modality completed second
  Interventions: Behavioral: Face-to-face evaluation (FF); Behavioral: TeleNP evaluation
- Care Partners (No Intervention): Care Partners did not undergo the intervention; they completed outcome measures (surveys) of acceptability only.

INTERVENTIONS:
Behavioral: Face-to-face evaluation (FF) — The intervention is the assessment modality. The control condition is face-to-face evaluation (FF).
  Arms: Face-to-face evaluation (FF), TeleNP evaluation; TeleNP evaluation, Face-to-face evaluation (FF)
Behavioral: TeleNP evaluation — The intervention is the assessment modality. The intervention condition is TeleNP evaluation.
  Arms: Face-to-face evaluation (FF), TeleNP evaluation; TeleNP evaluation, Face-to-face evaluation (FF)

SUMMARY:
The overarching goal of this study is to a) assess the feasibility and preliminary validity of home-based delivery of TeleNP to patients with suspected Alzheimer's Disease (AD), referred for cognitive assessments in a Neurology Clinic; and b) elucidate whether TeleNP is equivalent to face-to-face evaluation (FF) for diagnostic adjudication of atypical versus typical AD.

ELIGIBILITY:
Inclusion Criteria:

* Individuals age 60 to 90 years who are undergoing evaluation for possible AD and whose severity ranges from MCI to mild dementia.
* Individuals must carry a diagnosis of either suspected typical AD or atypical AD, based on the referring neurologist's diagnosis.

Exclusion Criteria:

* Individuals with moderate to severe levels of dementia and individuals with active delirium (per neurologist's determination).
* Individuals who are legally blind or deaf, due to the auditory and visual components of the study.
* Individuals with a brain tumor and individuals who have a confirmed nonAD neurological diagnosis (e.g, Multiple Sclerosis; FTD).
* Individuals who are being evaluated outside of the UCH Memory Disorders Clinic.
* Individuals who report active (i.e., within the last 6 months) substance use of illicit drugs such as cocaine or methamphetamines, or who carry a diagnosis of a major psychiatric disorder (e.g., schizophrenia; bipolar disorder).

Note that care partners (3rd arm) did not undergo the intervention and there were no additional eligibility requirements for them except that they were involved in the patient's care

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2022-06-27 (Actual); Primary Completion 2024-05-16 (Actual); Study Completion 2024-05-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brianne Bettcher, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus (CU-AMC), Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Intervention (Patients): Eligible participants were adults ≥age 60 years and <90 years whose severity was MCI or mild dementia. Behavioral neurologists referred patients based on: a) the patient was undergoing initial diagnostic evaluation, b) the neurologist intended to place a referral for a neuropsychological evaluation, and c) Alzheimer's Disease was on the differential diagnostic workup.
  Non-intervention (Care Partners): There were no eligibility requirements for the care partner
Pre-assignment Details: Intervention Arms (Patients): Upon consenting for the study, randomization was conducted using a computerized process through REDCap based on block randomization with blocks of sizes 32, 24, 16, and two of 8 based on modality (FF vs TeleNP) order, test form type (standard vs alternate; used for a subset of tests), and assigned to one of two board certified neuropsychologists.
  Non-Intervention Arm (Care Partner): Care partners were not assigned to an intervention, no pre-assignment details
Groups:
- Face-to-face Evaluation (FF), Teleneuropsychology Evaluation (TeleNP): Study participants underwent both modalities (FF; TeleNP), conducted 4-6 weeks apart (allowing for maximum of 90 days). Order of modality, either FF followed by TeleNP or vice versa, was randomized at baseline using a computerized process through REDCap.
- Teleneuropsychology Evaluation (TeleNP), Face-to-face Evaluation (FF): Study participants underwent both modalities (TeleNP; FF), conducted 4-6 weeks apart (allowing for maximum of 90 days). Order of modality, either TeleNP followed by FF or vice versa, was randomized at baseline using a computerized process through REDCap.
- Care Partners: Care partners of patients who were enrolled in the intervention trial were consented to fill out surveys. They did not undergo an intervention.
Period: Overall Study
Arm/Group | Face-to-face Evaluation (FF), Teleneuropsychology Evaluation (TeleNP) | Teleneuropsychology Evaluation (TeleNP), Face-to-face Evaluation (FF) | Care Partners
Started | 35 | 31 | 50
Completed | 32 | 31 | 50
Not Completed | 3 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The n=50 care partners did not undergo the intervention
Groups:
- Care Partner: Care Partners did not undergo the intervention. They filled out acceptability surveys, which were an outcome measure
- Total: Total of all reporting groups
Arm/Group | Face-to-face Evaluation (FF), Teleneuropsychology Evaluation (TeleNP) | Teleneuropsychology Evaluation (TeleNP), Face-to-face Evaluation (FF) | Care Partner | Total
Number analyzed (Participants) | 32 | 31 | 50 | 113
Age, Continuous [Mean (Standard Deviation); unit: Years] — Total column reflects intervention only metrics, and doesn't include care partners (who did not participate in an intervention) Population: Differences between numbers: 3 participants signed consent but did not complete baseline
  Years
    Patients: number analyzed (Participants) | 32 | 31 | 0 | 63
    Patients | 73.03 (6.49) | 73.74 (6.16) |  | 73.38 (6.29)
    Care Partners: number analyzed (Participants) | 0 | 0 | 50 | 50
    Care Partners |  |  | 63.8 (12.6) | 63.8 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Differences between numbers: 3 participants signed consent but did not complete baseline
  Participants
    Female | 15 | 20 | 33 | 68
    Male | 17 | 11 | 17 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Differences between numbers: 3 participants signed consent but did not complete baseline
  Participants
    Hispanic or Latino | 2 | 0 | 2 | 4
    Not Hispanic or Latino | 30 | 31 | 48 | 109
    Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Differences between numbers: 3 participants signed consent but did not complete baseline
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0
    Asian | 0 | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
    Black or African American | 1 | 1 | 2 | 4
    White | 30 | 29 | 47 | 106
    More than one race | 1 | 0 | 1 | 2
    Unknown or Not Reported | 0 | 0 | 0 | 0
Diagnosis (By Referring Neurologist): Atypical AD, Typical AD [Count of Participants; unit: Participants] — "Typical AD" was defined as patients with a memory-predominant presentation of AD. "Atypical/complex AD" was defined as patients with either a) a non-memory predominant phenotype of AD or b) a complex/unclear presentation Population: Differences between numbers: 3 participants signed consent but did not complete baseline
  Participants
    number analyzed (Participants) | 32 | 31 | 0 | 63
    Atypical AD | 12 | 10 | 0 | 22
    Typical AD | 20 | 21 | 0 | 41
Severity Level: MCI, Mild Dementia [Count of Participants; unit: Participants] — MCI and Dementia level of severity were based on neurologist determination, consistent with NIA-AA clinical criteria. MCI represents a change in cognitive functioning from baseline, with activities of daily living mostly preserved. Dementia represents a change in cognitive functioning from baseline that impacts activities of daily living. Dementia represents a greater/worse severity level than MCI. Population: Differences between numbers: 3 participants signed consent but did not complete baseline
  Participants
    number analyzed (Participants) | 32 | 31 | 0 | 63
    MCI | 24 | 22 | 0 | 46
    Mild Dementia | 8 | 9 | 0 | 17

OUTCOME MEASURES:

1. Primary Outcome: Agreement of Cognitive Test Results Across Testing Modalities as Measured by Neuropsychological Test Mean Scores, Measures With Total Correct Items
Description: Raw scores for measures of Memory, Executive Functions, Language, and Spatial Abilities will be compared across both conditions.
  CVLT= California Verbal Learning Test- 2nd edition; Delayed recall measures Memory, total words recalled after 20-minutes (range: 0-16). Higher=better.
  RBANS = Repeatable Battery for the Assessment of Neuropsychological Status; Delayed recall (Memory) - total elements recalled (range: 0-20). Higher=better.
  Figure Copy (Spatial)- total copied (range: 0-20). BNT=Boston Naming Test (Language) -total correct (range: 0-15). Higher=better. Category Fluency (Language) - total correct) (range: 0- no limit). Higher=better.
  JoLO=Judgment of Line Orientation (Spatial) -total correct (range: 0-15). Higher=better
Time Frame: After the exposure to each health delivery conditions, Face-to-face evaluation (FF) and TeleNP evaluation, at Week 1 and Weeks 5-7
Population: Three participants who underwent the intervention signed a consent but did not complete baseline. Care Partners did not undergo the intervention and thus are not included in these outcomes.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Teleneuropsychology (TeleNP): Neuropsychological assessment administered via remote, home-based telehealth
- Face-to-Face (FF): Neuropsychological assessment administered in-person
Arm/Group | Teleneuropsychology (TeleNP) | Face-to-Face (FF)
Number analyzed (Participants) | 63 | 63
score on a scale
  CVLT Delayed Recall (Memory). Total Score, Higher=better score. | 4.31 (4.30) | 4.40 (4.20)
  RBANS Figure Delayed Recall (Memory). Total Score, Higher=better score. | 8.21 (5.20) | 8.60 (4.90)
  BNT-15 item Total (Language), Total Score, Higher=better score. | 12.40 (3.20) | 12.52 (3.20)
  Category Fluency Total (Language), Total Score, Higher=better score. | 13.19 (5.50) | 12.83 (5.80)
  JoLO 15-item Total (Spatial), Total Score, Higher=better score. | 10.60 (3.40) | 11.10 (3.00)
  RBANS Figure Copy (Spatial), Total Score, Higher=better score. | 17.08 (2.50) | 17.21 (2.60)
Statistical Analysis 1: Comparison: Teleneuropsychology (TeleNP) vs Face-to-Face (FF); Unadjusted intraclass correlation coefficient (ICC) estimates and their 95% confidence intervals were calculated for each outcome measure to assess the reliability of measures across condition type based on a single-rating, absolute-agreement, two-way random-effects model. Results for Memory: CVLT shown below; Test type: Other — Intraclass correlation coefficient (ICC); ICC estimates and 95% CIs were interpreted as agreement across condition type, where estimates of 0-<0.50 are considered poor, 0.50≤-<0.75 moderate, 0.75≤-<0.90 good, and 0.90≤-1 excellent. ICCs were adjusted for age and sex; Not applicable, ICC level of agreements interpreted; IntraClassCorrelation = 0.67, 95% CI 2-sided [0.50 to 0.78] — ICC with 95% CI for Memory, CVLT delayed recall shown
Statistical Analysis 2: Comparison: Teleneuropsychology (TeleNP) vs Face-to-Face (FF); Unadjusted intraclass correlation coefficient (ICC) estimates and their 95% confidence intervals were calculated for each outcome measure to assess the reliability of measures across condition type based on a single-rating, absolute-agreement, two-way random-effects model. Results for Memory: RBANS shown below; Test type: Other — Intraclass correlation coefficient (ICC); [p-value comment as in outcome 1, analysis 1]; Not applicable, ICC level of agreements interpreted; Intraclass Correlation = 0.74, 95% CI 2-sided [0.71 to 0.84] — ICC with 95% CI for Memory, RBANS delayed recall shown
Statistical Analysis 3: Comparison: Teleneuropsychology (TeleNP) vs Face-to-Face (FF); Unadjusted intraclass correlation coefficient (ICC) estimates and their 95% confidence intervals were calculated for each outcome measure to assess the reliability of measures across condition type based on a single-rating, absolute-agreement, two-way random-effects model. Results for Memory: BNT-15 shown below; Test type: Other — Intraclass correlation coefficient (ICC); [p-value comment as in outcome 1, analysis 1]; Not applicable, ICC level of agreements interpreted; Intraclass correlation = 0.85, 95% CI 2-sided [0.76 to 0.90] — ICC with 95% CI for Language, BNT-15 shown
Statistical Analysis 4: Comparison: Teleneuropsychology (TeleNP) vs Face-to-Face (FF); Unadjusted intraclass correlation coefficient (ICC) estimates and their 95% confidence intervals were calculated for each outcome measure to assess the reliability of measures across condition type based on a single-rating, absolute-agreement, two-way random-effects model. Results for Lang8age: Category Fluency shown below; Test type: Other — Intraclass correlation coefficient (ICC); [p-value comment as in outcome 1, analysis 1]; Not applicable, ICC level of agreements interpreted; intraclass correlation = 0.76, 95% CI 2-sided [0.63 to 0.85] — ICC with 95% CI for Language, Category Fluency shown
Statistical Analysis 5: Comparison: Teleneuropsychology (TeleNP) vs Face-to-Face (FF); Unadjusted intraclass correlation coefficient (ICC) estimates and their 95% confidence intervals were calculated for each outcome measure to assess the reliability of measures across condition type based on a single-rating, absolute-agreement, two-way random-effects model. Results for Spatial: JoLO 15-item Total; Test type: Other — Intraclass correlation coefficient (ICC); [p-value comment as in outcome 1, analysis 1]; Not applicable, ICC level of agreements interpreted; Intraclass correlation = 0.62, 95% CI 2-sided [0.45 to 0.75] — ICC with 95% CI for Spatial, JoLO-15 item shown
Statistical Analysis 6: Comparison: Teleneuropsychology (TeleNP) vs Face-to-Face (FF); Unadjusted intraclass correlation coefficient (ICC) estimates and their 95% confidence intervals were calculated for each outcome measure to assess the reliability of measures across condition type based on a single-rating, absolute-agreement, two-way random-effects model. Results for Spatial: RBANS Figure Copy shown below; Test type: Other — Intraclass correlation; [p-value comment as in outcome 1, analysis 1]; Not applicable, ICC level of agreements interpreted; Intraclass correlation = 0.57, 95% CI 2-sided [0.38 to 0.72] — ICC with 95% CI for Spatial, RBANS Figure Copy shown

2. Primary Outcome: Agreement of Neuropsychologist Diagnosis Across Testing Modalities as Measured by Neuropsychologist-Determined Diagnosis
Description: Neuropsychologist-determined diagnosis (i.e., typical AD, atypical/complex AD, not AD) will be compared across both conditions whether TeleNP alters assessment of patient diagnosis.
Time Frame: as for outcome 1
Population: Three participants signed a consent but did not complete baseline. Neuropsychologist (n=2 neuropsychologists)-determine diagnostic agreement for all participants (n=63) will be determined between the modalities.
Measure: Mean (95% Confidence Interval); unit: Cohen's Kappa
Groups:
- Syndrome Across Modalities: Neuropsychologist Rating of Typical AD, Atypical AD, or not AD between TeleNP and FF
Arm/Group | Syndrome Across Modalities
Number analyzed (Participants) | 63
Cohen's Kappa | 0.74 [0.60 to 0.88]
Statistical Analysis 1: Comparison: Syndrome Across Modalities; We constructed 3x3 tables for the diagnostic considerations by core battery and syndrome impression by condition. Agreement between each question and impression category was determined using Cohen's kappa (unweighted). Kappa values were interpreted using the agreement categories as follows: 0-.20 as "None", .21-.39 as "Minimal", .40-.59; Test type: Other — Cohen's Kappa; Not applicable, Cohen's Kappa with level of agreement between neuropsychologists used; Cohen's Kappa = 0.74, 95% CI 2-sided [0.60 to 0.88]

3. Primary Outcome: Agreement of Neuropsychologist Appraisal of Severity Across Testing Modalities as Measured by Neuropsychologist-Determined Severity
Description: Neuropsychologist-determined severity (i.e., subjective cognitive concerns; MCI; mild dementia) will be compared across both conditions whether TeleNP alters assessment of patient severity.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: Cohen's Kappa
Groups:
- Severity Across Modalities: Neuropsychologist Rating of Subjective Concerns, MCI, and Dementia Across TeleNP and FF
Arm/Group | Severity Across Modalities
Number analyzed (Participants) | 63
Cohen's Kappa | 0.89 [0.79 to 0.99]
Statistical Analysis 1: Comparison: Severity Across Modalities; We constructed 3x3 tables for the diagnostic considerations by core battery and severity impression by condition. Agreement between each question and impression category was determined using Cohen's kappa (unweighted). Kappa values were interpreted using the agreement categories as follows: 0-.20 as "None", .21-.39 as "Minimal", .40-.59; Test type: Other — Cohen's Kappa; Not applicable, Cohen's Kappa with level of agreement between neuropsychologists used; Cohen's Kappa = 0.89, 95% CI 2-sided [0.79 to 0.99]

4. Primary Outcome: Acceptability and Feasibility of Intervention Measures as Measured by 4-item Acceptability and Feasibility of Intervention Measures Scale
Description: The 4-item Acceptability and Feasibility of Intervention Measures Scale is used for rating all participants and care partners' perspective on the acceptability and feasibility of the Face-to-face evaluation (FF) and TeleNP evaluation as assessed using a 5-point Likert scale at Week 1 or Weeks 5-7, depending on randomization. Scores range from "Completely disagree" (1) to "Completely agree" (5).
Time Frame: as for outcome 1
Population: For the patients (i.e., the primary participants), 3 participants signed a consent but did not complete baseline. N=63.
  For the care partners, it was not a requirement that the patient's have a care partner. Results are provided for the care partners who were available and consented (n=50).
Measure: Median (Inter-Quartile Range); unit: Score on a Scale
Groups:
- Patient (Acceptability Measure): Patient (primary participant) report of acceptability measures
- Care Partner (Acceptability Measure): Care Partner (care partner of primary participant/patient) report of acceptability measures
Arm/Group | Patient (Acceptability Measure) | Care Partner (Acceptability Measure)
Number analyzed (Participants) | 63 | 50
Score on a Scale
  TeleNP. Acceptability of Intervention Measure. Range 1-5; Higher=More Acceptable | 4.0 [3.5 to 4.5] | 3.95 [3.3 to 4.8]
  TeleNP. Intervention Appropriateness Measure. Range 1-5; Higher=More Acceptable | 4.0 [3.5 to 4.3] | 4.0 [3.5 to 4.5]
  TeleNP. Feasibility of Intervention Measure. Range 1-5; Higher=More Acceptable | 4.0 [3.8 to 4.5] | 4.0 [3.8 to 4.8]
  FF (Face-to-Face). Acceptability of Intervention Measure. Range 1-5; Higher=More Acceptable | 4.0 [3.5 to 5.0] | 3.9 [3.5 to 4.3]
  FF (Face-to-Face). Intervention Appropriateness Measure. Range 1-5; Higher=More Acceptable | 4.0 [4.0 to 4.8] | 4.0 [4.0 to 4.8]
  FF (Face-to-Face). Feasibility of Intervention Measure. Range 1-5; Higher=More Acceptable | 4.0 [3.8 to 4.8] | 4.0 [3.8 to 4.8]

5. Primary Outcome: Acceptability and Feasibility of Intervention Measures as Measured by 19-item UTAUT Questionnaire Adapted to TeleNP
Description: The UTAUT questionnaire adapted to TeleNP is used for rating all participants' perspective on the acceptability and feasibility of TeleNP evaluation as assessed using a 5-point Likert scale at Week 1 or Weeks 5-7, depending on randomization. Scores range from "Strongly disagree" (1) to "Strongly agree" (5).
  Performance expectancy refers to the degree to which an individual believes that using a technology will help them improve their performance.
  Effort expectancy is the degree of ease associated with using the technology. Behavioral intention reflects an individual's plan to use the technology.
Time Frame: After the exposure to the TeleNP evaluation (up to Week 7)
Population: For the patients (i.e., the primary participants), 3 participants signed a consent but did not complete baseline. N=63.
Measure: Median (Full Range); unit: Score (Higher=more acceptable, range 1-5
Groups:
- Patient (UTAUT Measure): Patient (primary participant) report on UTAUT measure
Arm/Group | Patient (UTAUT Measure)
Number analyzed (Participants) | 63
Score (Higher=more acceptable, range 1-5
  Performance Expectancy Domain | 4.0 [3.0 to 5.0]
  Effort Expectancy Domain | 4.0 [3.0 to 4.0]
  Behavioral Intention Domain | 4.0 [3.0 to 4.0]

6. Primary Outcome: Agreement of Cognitive Test Results Across Testing Modalities as Measured by Neuropsychological Test Mean Scores (Timed Measures)
Description: Raw scores for measures of Executive Functions will be compared across both conditions.
  DKEFS= Delis-Kaplan Executive Function Systems; Color-Word Inhibition (Executive Functions) -total time (range: 0-180"). Higher=worse Oral Trail Making Test B (Executive Functions) total time (range: 0-300"). Higher=worse
Time Frame: as for outcome 1
Population: Three participants signed a consent but did not complete baseline
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Teleneuropsychology (TeleNP) | Face-to-Face (FF)
Number analyzed (Participants) | 63 | 63
seconds
  DKEFS Color-Word Inhibition Total Time | 104.84 (44.10) | 96.29 (38.10)
  Oral Trail Making Test, Total Time | 88.54 (87.10) | 79.59 (83.30)
Statistical Analysis 1: Comparison: Teleneuropsychology (TeleNP) vs Face-to-Face (FF); Unadjusted intraclass correlation coefficient (ICC) estimates and their 95% confidence intervals were calculated for each outcome measure to assess the reliability of measures across condition type based on a single-rating, absolute-agreement, two-way random-effects model. Results for Executive Functions: DKEFS Color Word Inhibition shown below; Test type: Other — Intraclass correlation coefficient (ICC); [p-value comment as in outcome 1, analysis 1]; Not applicable, ICC level of agreements interpreted; Intraclass correlation = 0.82, 95% CI 2-sided [0.71 to 0.89] — ICC with 95% CI for Executive Functions, DKEFS Color Word-Inhibition shown
Statistical Analysis 2: Comparison: Teleneuropsychology (TeleNP) vs Face-to-Face (FF); Unadjusted intraclass correlation coefficient (ICC) estimates and their 95% confidence intervals were calculated for each outcome measure to assess the reliability of measures across condition type based on a single-rating, absolute-agreement, two-way random-effects model. Results for Executive Functions:Oral Trail Making Test B shown below; Test type: Other — Intraclass correlation coefficient (ICC); [p-value comment as in outcome 1, analysis 1]; Not applicable, ICC level of agreements interpreted; Intraclass correlation = 0.88, 95% CI 2-sided [0.81 to 0.93] — ICC with 95% CI for Executive Functions, Oral Trail Making Test B shown

ADVERSE EVENTS:
Time Frame: From enrollment until the patient's evaluation feedback session (i.e., when final feedback session was conducted to the patient, within 3 months of their baseline visit). Note that care partners (arm 3) did not undergo the intervention and thus AEs were not collected or reported.
Description: Note that care partners (arm 3) did not undergo the intervention and thus AEs were not collected or reported.
Groups:
- Face-to-face Evaluation (FF): Face to Face evaluation (standard of care)
- Teleneuropsychology Evaluation (TeleNP): Teleneuropsychology evaluation, intervention condition
Arm/Group | Face-to-face Evaluation (FF) | Teleneuropsychology Evaluation (TeleNP)
All-Cause Mortality (participants affected / at risk) | 0/63 | 0/63
Serious Adverse Events (participants affected / at risk) | 0/63 | 0/63
Other Adverse Events (participants affected / at risk) | 0/63 | 0/63

LIMITATIONS AND CAVEATS:
* Our trial sample size was relatively small and our sample was lacking in racial/ethnic diversity.
* The division of syndromes into three categories (typical AD; atypical AD; not AD) does not map onto NIA-AA diagnostic criteria which require both clinical diagnoses and biomarker evaluation of AD pathology; however, most neuropsychologists do not have access to biomarkers in clinical practice.
* Standardization of patients' home environment remains a challenge.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-11): https://cdn.clinicaltrials.gov/large-docs/23/NCT05379023/Prot_SAP_000.pdf